CLINICAL TRIAL: NCT04101448
Title: Prevalence of and Prognostic Impact of Bronchiectasis in COPD Patients
Brief Title: Prevalence of Bronchiectasis in COPD Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aliae AR Mohamed Hussein, Professor of Pulmonology, Assiut University
Other Study IDs: AssiutU7
Record Dates: First submitted 2019-09-22; First posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Bronchiectasis; Chronic Obstruct Airways Disease; Prognosis
Keywords: Bronchiectasis; COPD; Prevalence; Prognosis
MeSH Terms: conditions — Bronchiectasis; Pulmonary Disease, Chronic Obstructive | interventions — Prevalence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: COPD patients with bronchiectasis
  Interventions: Other: prevalence
- Group B: COPD patients without bronchiectasis
  Interventions: Other: prevalence

INTERVENTIONS:
Other: prevalence — percentage of bronchectasis in COPD and its effect as prognostic measure

SUMMARY:
The identification of bronchiectasis in COPD has been defined as a different clinical COPD phenotype with greater symptomatic severity, more frequent chronic bronchial infection and exacerbations, and poor prognosis. A causal association has not yet been proven, but it is biologically plausible that COPD, and particularly the infective and exacerbator COPD phenotypes, could be the cause of bronchiectasis without any other known etiology, beyond any mere association or comorbidity.

DETAILED DESCRIPTION:
The relationship between bronchiectasis and COPD has generated several questions. Is there any real increased prevalence of bronchiectasis in patients with COPD? Does the presence of bronchiectasis have an impact on the clinical characteristics, prognosis, or response to treatment in COPD, to the extent that it can be considered a distinct clinical phenotype? Should bronchiectasis in patients with COPD be seen as merely a comorbidity, or as a consequence of the disease's natural history? Is there a causal relationship between COPD and bronchiectasis? If this is the case, what are the pathophysiological mechanisms responsible for this relationship? And, finally, what is the role of chronic bronchial infection and exacerbations in this relationship?

ELIGIBILITY:
Inclusion Criteria:

* COPD patients based on GOLD 2019 criteria, stable or in exacerbation

Exclusion Criteria:

* acute pneumonia within 2 months
* malignancy
* congenital bronchiectasis ( immobile cilia syndrome, Kartagnar syndrome).
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: COPD patients diagnosed based on GOLD criteria 2019 with chest CT finding of bronchiectasis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-09-30 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Bronchiectasis in COPD | 1 year
  percentage of bronchiectasis diagnosed by CT chest in COPD patients

SECONDARY OUTCOMES:
impact of bronchiectasis on COPD exacerbations | 1 year
  number of exacerbations treated in or out of hospitals
impact of bronchiectasis on COPD hospitalization | 1 year
  number of hospital admissions with acute exacerbations
impact of bronchiectasis on COPD intensive care admission | 1 year
  number of admissions in respiratory ICU and need for mechanical or non invasive ventilation

CONTACTS AND LOCATIONS:
Locations (1):
- AssiutU, Asyut, Egypt